CLINICAL TRIAL: NCT05176288
Title: Avelumab, Palbociclib and Axitinib in in Treatment Naive Metastatic Clear Cell Renal Cell Carcinoma.
Brief Title: Avelumab, Palbociclib and Axitinib in Advanced RCC
Acronym: APART
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The overall protocol will be changed in a new amendment, which will be resubmitted under the new IND.
Sponsor: Bradley A. McGregor, MD (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Bradley A. McGregor, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-575
Record Dates: First submitted 2021-12-06; First posted 2022-01-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma
Keywords: Advanced Clear Cell Renal Cell Carcinoma
MeSH Terms: interventions — Axitinib; palbociclib; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axitinib, Avelumab and Palbociclib (Experimental): During each 28 day (+/- 3 days) study cycle, all participants will receive:
  * Axitinib: 2x Daily until it is determined participant must stop the drug
  * Palbociclib: Taken 1x time per day on days 8-28 of each cycle until it is determined participant must stop the drug.
  * Avelumab: Once every 2 weeks continued for up to 2 years or earlier if it is determined participant must stop the study drug
  Interventions: Drug: Axitinib; Drug: Palbociclib; Drug: Avelumab

INTERVENTIONS:
Drug: Axitinib — Taken Orally
  Other Names: Inlyta
Drug: Palbociclib — Taken Orally
  Other Names: Ibrance
Drug: Avelumab — Intravenous infusion
  Other Names: Bavencio

SUMMARY:
The aim of this study is to see whether the combination of 3 drugs (axitinib, avelumab and palbociclib) is safe and effective in slowing down the growth of advanced clear cell renal cell carcinoma (ccRCC) in patients that have not received any prior systemic treatment.

The names of the study drug involved in this study are/is:

* Axitinib
* Avelumab
* Palbociclib

DETAILED DESCRIPTION:
This is a multi-center, single-arm, phase 2 study to evaluate the efficacy of the combination of axitinib, avelumab, and palbociclib in patients with untreated, advanced clear cell renal cell carcinoma (ccRCC).

This research study involves an investigational drug combination (axitinib, avelumab and palbociclib) not approved by the FDA (USA Food and Drug Administration) for treatment of advanced clear cell renal cell carcinoma (ccRCC), though the combination of axitinib and avelumab has been approved for use in advanced clear cell renal cell carcinoma (ccRCC) treatment. Palbociclib is a CDK inhibitor, which targets growing cancer cells by blocking how a phosphate molecule is added to an important regulatory protein called retinoblastoma so preventing the formation of new cancer cells.

Study procedures include screening for eligibility, study treatment, participant evaluations and safety follow visits in addition to general health status follow-up after study treatment. Participants will receive study treatment for as long as they do not have serious side effects and their disease does not get worse, and will be followed for as long as they remain on the study.

It is expected that about 25 people will take part in this research study.

Pfizer is supporting this research study by providing the study drugs (axitinib, avelumab and palbociclib).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable advanced or metastatic renal cell carcinoma with a clear cell component. Patient with sarcomatoid histology are accepted.

  * A formalin-fixed, paraffin-embedded (FFPE) tumor tissue block from a de novo tumor biopsy obtained during screening will be required (biopsied tumor lesion should not be a RECIST target lesion). Alternatively, a recently obtained archival FFPE tumor tissue block (not cut slides from a primary or metastatic tumor resection or biopsy) can be provided if the following criteria are met:

    * The biopsy or resection was performed within 1 year of registration AND
    * The patient has not received any intervening systemic anti-cancer treatment from the time the tissue was obtained and registration onto the current study. If an FFPE tissue block cannot be provided as per documented regulations then 15 unstained slides (10 minimum) will be acceptable
  * Availability of an archival FFPE tumor tissue block from primary diagnosis specimen (if available and not provided per above). If an FFPE tissue block cannot be provided as per documented regulations, then 15 unstained slides (10 minimum) will be acceptable
  * Additional tumor biopsies for research purposes prior to starting therapy, after 2 months of therapy and at end of treatment are optional.
* Measurable disease as per RECIST 1.1. See section 11 for the evaluation of measurable disease.
* Age ≥ 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1.5×109/L
  * Platelets ≥100×109/L
  * Hemoglobin ≥9g/dL (transfusions allowed)
  * Total bilirubin ≤2 × institutional upper limit of normal (ULN) with the following exception: patients with known Gilbert disease should have a serum bilirubin ≤ 3 x ULN
  * AST(SGOT)/ALT(SGPT) ≤3 × ULN with the following exception: patients with known liver metastases should have AST and ALT ≤ 5 × ULN
  * Creatinine clearance ≥30 mL/min according to the Cockcroft-Gault equation. (APPENDIX F)
  * Urine protein <2+ by dipstick; if dipstick ≥2+, then 24 hour urinary protein <2g
* Women of child-bearing potential and men must agree to use adequate contraception (intrauterine device or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. A negative pregnancy serum test should be obtained within 7 days of therapy initiation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation. Participants treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 30 days after completion of avelumab, axitinib and palbociclib administration.
* Ability to swallow oral medications.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Treatment with the following prior therapies:

  * Prior systemic therapy for advanced or metastatic RCC.
  * Prior adjuvant or neoadjuvant therapy for RCC if disease progression or relapse has occurred within 12 months of last dose of such therapy. Treatment with an immune checkpoint inhibitor in the adjuvant setting is allowed providing more than 12 months have elapsed since completion of therapy.
  * Prior treatment with any immunotherapeutic agent (IL-2, IFN-∝, anti-PD(L)-1, anti-CTLA-4, or any other antibody or drug targeting T-cell co-stimulation or immune checkpoint pathways).
  * Prior therapy with axitinib or other therapies targeting VEGF pathway in the metastatic setting (adjuvant therapy is allowed.
  * Prior therapy with any CDK4/6 inhibitor.
* Participants with untreated brain metastases. Participants with metastatic CNS tumors may participate in this trial, if the participant is ≥ 4 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy >10 mg/day prednisone or equivalent. A repeat MRI or CT brain to show stability is required.
* Participants who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy to at least grade 1.
* Untreated deep vein thrombosis or pulmonary embolism, or event of deep vein thrombosis or pulmonary embolism within 2 weeks of treatment start. Patient should be on at least 1 week of anticoagulation before C1D1.
* Major surgery within the past 4 weeks or major radiation therapy within 2 weeks prior to treatment start. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed at least 48 hours prior to patient randomization.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease - also see 3.2.22, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Persisting toxicity related to prior therapy NCI CTCAE v5.0 Grade >1; however, sensory neuropathy Grade ≤2 is acceptable.
* Current or prior use of immunosuppressive medication within 7 days prior to randomization, except the following:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg. intra-articular injection).
  * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent.
  * Steroids as premedication for hypersensitivity reactions (eg. CT scan premedication).
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade≤3) or any history of anaphylaxis.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines).
* Grade≥3 hemorrhage within 4 weeks of registration
* Patient with active systemic bacterial infection (requiring IV antibiotics at the time of initiating study treatment), fungal infection, or detectable viral infection. Patients with known viral infection (such as HIV) are excluded given the potential for interactions between antiretroviral agents and palbociclib and axitinib, and the potential for increased risk of life-threatening infection with therapy that is myelosuppressive. If patients are not known to have HIV, a HIV test is required.
* Patients with known Hepatitis B or Hepatitis C infection are excluded only if there is evidence of active infection (detectable Hepatitis B surface antigen, detectable Hepatitis C RNA).
* Prior allogenic stem cell or solid organ transplant.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Participants who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant. Therapeutic use of low molecular weight heparin and factor Xa inhibitors (eg. apixaban, rivaroxaban) is permitted.
* Other malignancy diagnosed within 2 years of treatment start unless negligible risk of metastases or death according to the investigator (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma, or other malignancy not deemed to impact patients 5-year life expectancy).
* Has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), sudden cardiac arrest.
* Has had any major cardiovascular event within 6 months prior to treatment start, including but not limited to: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic event or New York Heart Association Class III or IV heart failure.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2 or prolongation of the QTc interval to >500 msec.
* History of interstitial lung disease or other restrictive lung disease, as well as history of symptomatic respiratory condition considered clinically significant by the investigator. Individuals with a history of radiotherapy to the thorax will be excluded.
* Active or ex-smokers with a history of cigarette smoking greater than 30pack-yrs (i.e., # of packs of cigarettes smoked per day x # of years patient has smoked > 30).
* Participants with a known hypersensitivity to the study compounds or to its excipients.
* Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors, including their administration within 10 days prior to treatment start (eg. grapefruit juice or grapefruit/grapefruit-related citrus fruits [eg. Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
* Current use or anticipated need for drugs that are known strong CYP3A4/5 inducers, including their administration within 10 days prior to treatment start (eg. phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St John's wort).
* Participants who have taken herbal medications within 7 days prior to treatment start. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
* Females that are pregnant or lactating.
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, for duration of therapy assessed up to 100 months
  Objective response rate (ORR) is defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taken as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.

SECONDARY OUTCOMES:
Median Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Based on the Kaplan-Meier method, median progression-free survival (PFS) is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of the longest diameter (LD) of target lesions taken as reference of the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Disease progression (PD) for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Median Overall Survival (OS) | Participants followed for long-term for survival every 6 months from the end of treatment until death or lost to follow-up, up to 2 years after treatment discontinuation.
  Based on the Kaplan-Meier method overall survival (OS) is defined as the time from study entry to death or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu